CLINICAL TRIAL: NCT04694300
Title: Demonstration of OTC Naproxen Sodium's (Aleve's) Anti-inflammatory Action in Dental Implant Surgery Patients
Brief Title: OTC Naproxen and Acetaminophen Anti-Inflammatory Action in Dental Implant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hersh, Elliot V., DMD, MS, PhD (Individual)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 844440; IIR (Other Grant/Funding Number: Bayer Pharmaceutical)
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Osseointegrated Dental Implantation; Pain, Acute
Keywords: Naproxen sodium; Acetaminophen; Postsurgical dental pain; Prostaglandins; Interleukins
MeSH Terms: conditions — Acute Pain | interventions — Naproxen; Acetaminophen; Tramadol

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, active-controlled, two arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Administration of naproxen or acetaminophen will be masked by over-encapsulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naproxen sodium (Experimental): Naproxen sodium 440 mg followed by naproxen sodium 220 mg q 8h (max 660 mg/day)
  Interventions: Drug: Naproxen; Drug: Tramadol
- Acetaminophen (Active Comparator): Acetaminophen 1000 mg followed by acetaminophen 1000 mg q 6h (max 3000 mg/day according to Tylenol package insert)
  Interventions: Drug: Acetaminophen; Drug: Tramadol

INTERVENTIONS:
Drug: Naproxen — 440 mg by mouth immediately after completion of implant surgery followed by 220 mg 12 hours later.
  Then 220 mg every 8 hours for the next two days.
  Other Names: Aleve
  Arms: Naproxen sodium
Drug: Acetaminophen — 1000 mg by mouth immediately after the completion of implant surgery followed by 1000 mg every 6 hours for 3 days after surgery with a maximum daily dose of 3000 mg.
  Other Names: Extra Strength Tylenol
  Arms: Acetaminophen
Drug: Tramadol — 50 mg by mouth every 6 hours as needed for pain
  Other Names: Ultram

SUMMARY:
This double-blind pilot study will evaluate the anti-inflammatory and analgesic effects of an over-the-counter (OTC) regimen of naproxen sodium versus acetaminophen in patients receiving one or two (adjacent) dental implants. It will also confirm that naproxen sodium in the OTC dosage range is a good alternative to immediate-release opioid formulations, which are subject to misuse, abuse and diversion in this patient population.

DETAILED DESCRIPTION:
Placement of dental implants is a frequently performed outpatient surgical procedure, with United States dentists currently placing implants in approximately 500,000 patients per year.This procedure has become the gold standard for replacing missing teeth due to its high level of predictability and patient acceptance, with long-term success rates greater than 95%. Thus, the number of patients opting for this procedure over dentures and fixed bridges continues to increase. In the period between 1999 and 2000 only 0.7% of the USA population had missing teeth with implants in contrast to 5.7% between 2015 and 2016 It is estimated that by 2026, if the current pace of dental implant placement continues, approximately 17% of the population will have dental implants.

Dental implant surgery involves the incision of gingival tissue to expose the underlying bone, followed by the creation of a precise bony cavity where the implant will be placed using a specialized surgical drill, and lastly the screwing of the implant into bone using a specialized handpiece Thus, it is not surprising that post-surgical pain is a common sequela following dental implant surgery. Patients often experience post-surgical pain for several days after the placement of one to three dental implants, but at a pain intensity level that is generally less than that of dental impaction surgery. This post-surgical pain is inflammatory in nature; thus, NSAIDs have demonstrated efficacy and are the preferred analgesics in this patient population. Postoperative administration of intranasal ketorolac (SPRIX®) and oral acetaminophen 325 mg plus codeine 30 mg have both demonstrated efficacy.

The soft tissue and bony trauma associated with dental implant surgery upregulates inflammatory mediators both locally and systemically. Elevated levels of interleukin (IL)-6, IL-8, and macrophage inflammatory protein (MIP)-1β have been observed in gingival crevicular fluid (GCF) from the implant site and the adjacent teeth one week after surgery. Prostaglandin E2 has been measured in the GCF of teeth surrounding implant sites employing similar methodology. Additionally, standard periodontal flap and bony recontouring surgery, which shares many similarities to dental implant surgery, induces an upregulation in immunoreactive prostaglandin E2 and leukotriene B4 levels at the surgical site. Dental implant surgery also increases cytokine levels in plasma, indicative of a systemic inflammatory response. Thus, in addition to being a model to study the efficacy and tolerability of OTC analgesics, dental implant surgery also appears to be an excellent model to study the anti-inflammatory properties of NSAIDs such as naproxen sodium.

Therefore, the investigators propose to initiate a double-blind, pilot study to evaluate the anti-inflammatory and analgesic effects of an OTC regimen of naproxen sodium versus acetaminophen in dental implant surgery patients. Notably, the vast majority of these patients are over the age of 45, a patient demographic that is rarely captured in postsurgical dental pain studies. Compared to dental impaction surgery patients, implant surgery patients possess more comorbidities such as hypertension, hyperlipidemia and hyperglycemia Thus, while dental impaction patients are typically on few if any drugs, polypharmacy is more of the norm in dental implant surgery patients. Performing a controlled study with OTC naproxen sodium in this population will provide the opportunity to confirm that its short-term use is generally safe and effective in these older, more medically complex patients. It will also confirm that naproxen sodium in the OTC dosage range is a good alternative to immediate-release opioid formulations, which are subject to misuse, abuse and diversion in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires surgical placement of one or two (adjacent) dental implants
* Ability to read and sign informed consent
* Males and females for 18-75 years of age
* Non-smokers
* Negative urine drug screen

Exclusion Criteria

* Advanced periodontal disease (>20% Clinical Attachment Loss >20% radiographic bone loss)
* History of bisphosphonate usage
* Medical history or medical condition that makes any of the study medications (naproxen sodium, acetaminophen, tramadol, etc.) inappropriate treatment options including any scheduled or recent cardiac procedures (within 6 months), a history of GI ulcers, liver or kidney disease, and anticoagulant or lithium intake.
* History of an allergic reaction to any pain reliever/fever reducer
* Contraindication to opioid use
* Positive urine drug screen for drugs of abuse unless on stable doses of a non-analgesic drug for a legitimate medical purpose
* Pregnancy - A urine pregnancy test will be performed immediately before the scheduled surgery on all women of child-bearing potential
* Local or systemic diseases that affects wound healing and inflammatory biomarkers (diabetes, autoimmune (rheumatoid arthritis), or inflammatory disorders - osteoarthritis is allowed).
* Smokers on this pilot study because it can affect levels of inflammatory biomarkers - a urine cotinine test will be performed immediately prior to the scheduled surgery on all subjects even if participant denies smoking history
* History of systemic steroid use over 2 weeks within last 2 years.
* Poor oral hygiene on a non-compliant individual.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot V Hersh, DMD, MS, PhD, Principal Investigator — University of Pennsylvania; Katherine N Theken, PharmD, PhD, Principal Investigator — University of Pennsylvania School of Dental Medicine and Medicine
Locations (1):
- University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. This is a pilot, exploratory study.

REFERENCES:
- [Background] Moore PA, Hersh EV. Combining ibuprofen and acetaminophen for acute pain management after third-molar extractions: translating clinical research to dental practice. J Am Dent Assoc. 2013 Aug;144(8):898-908. doi: 10.14219/jada.archive.2013.0207. PMID 23904576
- [Background] Hersh EV, Moore PA, Grosser T, Polomano RC, Farrar JT, Saraghi M, Juska SA, Mitchell CH, Theken KN. Nonsteroidal Anti-Inflammatory Drugs and Opioids in Postsurgical Dental Pain. J Dent Res. 2020 Jul;99(7):777-786. doi: 10.1177/0022034520914254. Epub 2020 Apr 14. PMID 32286125
- [Background] Deeb GR, Deeb JG, Agarwal V, Laskin DM. Use of transalveolar sutures to maintain vestibular depth and manipulate keratinized tissue following alveolar ridge reduction and implant placement for mandibular prosthesis. J Oral Maxillofac Surg. 2015 Jan;73(1):48-52. doi: 10.1016/j.joms.2014.07.022. Epub 2014 Jul 30. PMID 25315314
- [Background] Schmitt A, Zarb GA. The longitudinal clinical effectiveness of osseointegrated dental implants for single-tooth replacement. Int J Prosthodont. 1993 Mar-Apr;6(2):197-202. PMID 8329098
- [Background] Zarb GA, Schmitt A. The longitudinal clinical effectiveness of osseointegrated dental implants in posterior partially edentulous patients. Int J Prosthodont. 1993 Mar-Apr;6(2):189-96. PMID 8329097
- [Background] Elani HW, Starr JR, Da Silva JD, Gallucci GO. Trends in Dental Implant Use in the U.S., 1999-2016, and Projections to 2026. J Dent Res. 2018 Dec;97(13):1424-1430. doi: 10.1177/0022034518792567. Epub 2018 Aug 3. PMID 30075090
- [Background] Bockow R, Korostoff J, Pinto A, Hutcheson M, Secreto SA, Bodner L, Hersh EV. Characterization and treatment of postsurgical dental implant pain employing intranasal ketorolac. Compend Contin Educ Dent. 2013 Sep;34(8):570-6. PMID 24564610
- [Background] Alissa R, Sakka S, Oliver R, Horner K, Esposito M, Worthington HV, Coulthard P. Influence of ibuprofen on bone healing around dental implants: a randomised double-blind placebo-controlled clinical study. Eur J Oral Implantol. 2009 Autumn;2(3):185-99. PMID 20467629
- [Background] Hashem AA, Claffey NM, O'Connell B. Pain and anxiety following the placement of dental implants. Int J Oral Maxillofac Implants. 2006 Nov-Dec;21(6):943-50. PMID 17190305
- [Background] Al-Khabbaz AK, Griffin TJ, Al-Shammari KF. Assessment of pain associated with the surgical placement of dental implants. J Periodontol. 2007 Feb;78(2):239-46. doi: 10.1902/jop.2007.060032. PMID 17274712
- [Background] Samieirad S, Afrasiabi H, Tohidi E, Qolizade M, Shaban B, Hashemipour MA, Doaltian Shirvan I. Evaluation of caffeine versus codeine for pain and swelling management after implant surgeries: A triple blind clinical trial. J Craniomaxillofac Surg. 2017 Oct;45(10):1614-1621. doi: 10.1016/j.jcms.2017.06.014. Epub 2017 Jul 5. PMID 28864284
- [Background] Emecen-Huja P, Eubank TD, Shapiro V, Yildiz V, Tatakis DN, Leblebicioglu B. Peri-implant versus periodontal wound healing. J Clin Periodontol. 2013 Aug;40(8):816-24. doi: 10.1111/jcpe.12127. Epub 2013 Jun 18. PMID 23772674
- [Background] Aboyoussef H, Carter C, Jandinski JJ, Panagakos FS. Detection of prostaglandin E2 and matrix metalloproteinases in implant crevicular fluid. Int J Oral Maxillofac Implants. 1998 Sep-Oct;13(5):689-96. PMID 9796154
- [Background] O'Brien TP, Roszkowski MT, Wolff LF, Hinrichs JE, Hargreaves KM. Effect of a non-steroidal anti-inflammatory drug on tissue levels of immunoreactive prostaglandin E2, immunoreactive leukotriene, and pain after periodontal surgery. J Periodontol. 1996 Dec;67(12):1307-16. doi: 10.1902/jop.1996.67.12.1307. PMID 8997678
- [Background] Li S, Yang Y, Yu C, Yao Y, Wu Y, Qian L, Cheung CW. Dexmedetomidine Analgesia Effects in Patients Undergoing Dental Implant Surgery and Its Impact on Postoperative Inflammatory and Oxidative Stress. Oxid Med Cell Longev. 2015;2015:186736. doi: 10.1155/2015/186736. Epub 2015 Jun 15. PMID 26171113
- [Background] Pietruski JK, Pietruska MD, Stokowska W, Pattarelli GM. Serum levels of interleukin-1 (IL-1), interleukin-6 (IL-6) and interleukin-8 (IL-8) in patients treated with dental implants. Rocz Akad Med Bialymst. 2001;46:28-37. PMID 11780571
- [Background] Aghaloo T, Pi-Anfruns J, Moshaverinia A, Sim D, Grogan T, Hadaya D. The Effects of Systemic Diseases and Medications on Implant Osseointegration: A Systematic Review. Int J Oral Maxillofac Implants. 2019 Suppl;34:s35-s49. doi: 10.11607/jomi.19suppl.g3. PMID 31116832
- [Result] Theken KN, Chen M, Wall DL, Pham T, Secreto SA, Yoo TH, Rascon AN, Chang YC, Korostoff JM, Mitchell CH, Hersh EV. A randomized, double-blind pilot study of analgesic and anti-inflammatory effects of naproxen sodium and acetaminophen following dental implant placement surgery. Front Pharmacol. 2023 May 17;14:1199580. doi: 10.3389/fphar.2023.1199580. eCollection 2023. PMID 37266144
- See also: 17 Dental Implant Industry Statistics and Trends. — http://brandongaille.com/17-dental-implant-industry-statistics-and-trends/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects scheduled in University of Pennsylvania School of Dental Medicine Periodontics Clinic to receive the surgical placement of one or two dental implants.
Period: Overall Study
Arm/Group | Naproxen Sodium | Acetaminophen
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium | Acetaminophen | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (14.9) | 45.5 (14.2) | 46.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 10 | 14
  White | 8 | 3 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: BMI (kg/m^2)] | 25.2 (3.6) | 26.8 (4.3) | 26.0 (4.0)
Length of Surgery [Mean (Standard Deviation); unit: Minutes] — Implant surgery length from administration of local anesthetic to placement of last suture
  Minutes | 71.1 (35.8) | 85.5 (30.6) | 78.4 (33.7)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Scores on Numeric Pain Intensity Scale 0-6 Hours
Description: Median maximum pain intensity scores where 0 = no pain and 10 = worst possible pain
Time Frame: Up to 6 hours
Population: Medium Greatest Pain Intensity Scores from 0-6 hours Following Dosing With Naproxen Sodium or Acetaminophen
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Naproxen Sodium: Naproxen sodium 440 mg followed by naproxen sodium 220 mg q 8h (max 660 mg/day)
  Naproxen: 440 mg by mouth immediately after completion of implant surgery followed by 220 mg 12 hours later.
  Then 220 mg every 8 hours for the next two days.
  Tramadol: 50 mg by mouth every 6 hours as needed for pain
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
score on a scale | 1 [0 to 2.0] | 3 [2.0 to 7.0]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority — Lower the maximum pain intensity score the more effective the analgesic; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Pain Intensity Scores From 6 Through 72 Hours (Multi-dose Phase)
Description: Pain intensity scores where 0 = no pain and 10 = worst possible pain
Time Frame: 6-72 hours Post initial Dose
Population: Mean Pain Intensity Scores from 6-72 hours Following Around-the-Clock Dosing With Naproxen Sodium or Acetaminophen
Measure: Mean (Inter-Quartile Range); unit: units on pain intensity scale
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
units on pain intensity scale | 0.3 [0 to 0.6] | 1.7 [0.3 to 3.2]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Peak Plasma IL-6 Concentrations
Description: Plasma IL-6 concentrations 6 hours after treatment measured by ELISA
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
pg/ml | 6.5 [6.1 to 13.4] | 12.1 [6.7 to 30.0]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Plasma IL-6 Change From Baseline
Description: Percent change in plasma IL-6 levels at 6 hours after treatment relative to baseline
Time Frame: 6 hours post dose
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
percentage change from baseline | 276.9 [181.3 to 348.4] | 519.1 [262.6 to 1091]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rescue Analgesic Use
Description: Number of patients requiring opioid rescue medication (tramadol) during inpatient phase (0-6 hours) in each treatment group
Time Frame: 0-6 hours
Population: Number of patients in each treatment group requiring opioid rescue medication (tramadol) during inpatient phase (0-6 hours)
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
participants | 0 | 3

6. Secondary Outcome: Rescue Medication Use Outpatient Phase (6-72 Hours)
Description: Number of patients requiring opioid rescue medication during outpatient phase in both treatment groups
Time Frame: 6-72 hours
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
participants | 2 | 5

7. Secondary Outcome: Peak GCF IL-1β Levels
Description: Levels of IL-1β in gingival crevicular fluid measured at 24 hours after treatment
Time Frame: 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
pg/ml | 263 [110 to 1293] | 456 [243 to 1590]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: COX-1 Activity Percent of Baseline (Pre-surgery)
Description: Cyclooxygenase (COX)-1 activity was evaluated ex vivo by quantifying serum thromboxane B2 levels
Time Frame: 6 hours post dose
Measure: Median (Inter-Quartile Range); unit: percentage of baseline blood levels
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
percentage of baseline blood levels | 3.7 [2.8 to 11.3] | 77.4 [44.2 to 84.0]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: COX-2 Activity
Description: COX-2 activity was evaluated ex vivo by quantifying plasma prostaglandin (PG)E2 levels following lipopolysaccharide (LPS) stimulation in whole blood,
Time Frame: 6 hours post-dose
Population: Patient in each group surgically receiving one or two implants
Measure: Median (Inter-Quartile Range); unit: percentage of baseline blood levels
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
percentage of baseline blood levels | 48.4 [20.3 to 113.7] | 52.4 [27.7 to 146.3]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney); Higher percentage inhibition relates to greater selectivity for COX-2

10. Secondary Outcome: Peak GCF IL-8levels
Description: Levels of IL-8 in gingival crevicular fluid measured at 24 hours after treatment
Time Frame: 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 15 | 15
pg/ml | 2962 [657 to 7976] | 5729 [1972 to 9119]
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: One week
Description: Does not differ from clinicaltrials.gov
Arm/Group | Naproxen Sodium | Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium (N=15) | Acetaminophen (N=15)
Headache (General disorders) | 1 (1) | 0 (0) — Occurred during outpatient dosing with naproxen sodium
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) — Patient felt on edge during in patient period after initial dose of acetaminophen 1000 mg.
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — One patient after 1st dose, one patient as outpatient (multidose phase)
emesis (Gastrointestinal disorders) | 0 (0) | 2 (2) — Vomiting one episode each. One patient during as inpatient after first dose and one patient as outpatient during multi-dose phase

LIMITATIONS AND CAVEATS:
Research study as described in the results manuscript only evaluated 30 subjects but it is the first of it's kind. Our analysis was not powered to comprehensively evaluate the clinical and demographic factors that influence the local and systemic inflammatory response to implant placement surgery or drug response. In addition, we excluded smokers and patients with diabetes, autoimmune diseases, or other comorbidities that might influence the inflammatory response to implant placement surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT04694300/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04694300/ICF_002.pdf